CLINICAL TRIAL: NCT05494515
Title: Enhancing Early Swallowing Recovery of Postoperative Rehabilitation Program in Older Patients With Subjective Dysphagia After Anterior Cervical Spine Surgery: a Randomized Controlled Trial
Brief Title: Enhancing Early Swallowing Recovery in Older Dysphagic Patients Afetr Anterior Cervical Spine Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 202206073RINB
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Hypopharyngeal Pressure Changes Between Before and After Swallowing Rehabiliation

STUDY DESIGN:
Intervention Model Description: two groups, the early swallowing rehabilitation program, or the routine care group
Who Masked: Participant, Care Provider, Investigator
Masking Description: participants in the routine care group would still receive the swallowing education.
  Care providior and investigator did not know what groups do the patients belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the early swallowing rehabilitation program (Experimental): swallowing problem eveluated by high resolution impedance manometry (HRIM). The early swallowing rehabilitation program based on the results of HRIM evaluation
  Interventions: Procedure: the early swallowing rehabilitation program
- the routine care group (No Intervention): patients recieve swallowing education

INTERVENTIONS:
Procedure: the early swallowing rehabilitation program — the early swallowing rehabilitation program based on the HRIM evaluation
  Arms: the early swallowing rehabilitation program

SUMMARY:
The early swallowing rehabilitation program in older patients receiving elective surgery is regarded to enhance the recovery pf swallowing ability. However, objective evidence of changes in swallowing in older patients after ACSS, or the effect of the early rehabilitation program on recovery, is limited.

The aim of this study is that changes in hypopharyngeal muscle after ACSS will be significantly higher in older patients who underwent rehabilitation program than those who did not go through the rehabilitation program. Postoperative pulmonary complications and mortality will be followed up until 5 weeks after ACSS.

DETAILED DESCRIPTION:
Backgrounds: The number of aging patients is increasing. Aging is associated with an increased risk of dysphagia because of cerebral atrophy, deterioration in nerve function, and a region-dependent decline in muscle mass, which affects the swallowing mechanism. During the anterior approach cervical spine (ACSS) surgery, the upper esophageal sphincter (UES) and pharyngeal muscle group, especially the hypopharynx, is suspended to allow the surgeon to approach the cervical disc. The patients have an increased risk of dysphagia because traction injury of the UES and the muscle groups of the hypopharynx is unavoidable. The early swallowing rehabilitation program in older patients receiving elective surgery is regarded to enhance the recovery pf swallowing ability. However, objective evidence of changes in swallowing in older patients after ACSS, or the effect of the early rehabilitation program on recovery, is limited.

High resolution impedance manometry (HRIM) has been developed and used for the evaluation of dysphagia. HRIM involves multiple pressure sensors that detect changes in impedance as the food bolus is transmitted through the pharyngeal region. Eating Assessment Tool (EAT-10) is the most frequently used questionnaire for screening dysphagia, where score ≥4 is abnormal. Most previous studies used subjective questionnaire to investigate changes in perioperative swallowing after ACSS. One study that used HRIM to evaluate perioperative swallowing changes in ACSS patients found a decrease in muscle strength in the hypopharyngeal muscle groups. However, the study only recruited fourteen patients, and the mean age of the patients was 59 years old.

Aim and hypothesis: Investigators aim to investigate whether early swallowing rehabilitation can be used to enhance the hypopharyngeal muscle recovery after ACSS in aged patients with subjective dysphagia (EAT-10 score ≥4). The hypothesis is that changes in hypopharyngeal muscle after ACSS will be significantly higher in older patients who underwent rehabilitation program than those who did not go through the rehabilitation program. Postoperative pulmonary complications and mortality will be followed up until 5 weeks after ACSS.

Methods: Fifteen patients aged 60 to 80 years who underwent elective ACSS surgery will be recruited. All patients will have their HRIM measurement taken and answer the EAT-10 questionnaire before surgery. One week after ACSS, patients with EAT-10 scores≥4 will have their HRIM measurements taken and be randomized into either the intervention group, who will be enrolled in the early swallowing rehabilitation program, or the routine care group. The patients in the intervention group will return to the rehabilitation clinic after participating in the rehabilitation program for two weeks, during which their compliance will be monitored by daily phone reminders with a speech therapist or research assistant. After four weeks of participating in the rehabilitation program (i.e. five weeks after surgery), all patients in both the intervention and routine care groups will have their HRIM measurement taken and answer the EAT-10 questionnaire again. Postoperative pneumonia and mortality were followed up until five weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 60 to 80 years who underwent elective ACSS surgery
* One week after ACSS, patients with EAT-10 scores≥4

Exclusion Criteria:

* patients have major organ dysfunction, such as hemodialysis

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2027-08-22 (Estimated); Study Completion 2028-08-22 (Estimated)

PRIMARY OUTCOMES:
The difference in pre-and postoperative hypopharyngeal pressure | preoperative condition to postoperative 5 weeks

IPD SHARING:
Plan to Share IPD: No
due to ethical issue